CLINICAL TRIAL: NCT05738018
Title: An Observational Study Analyzing Patient Experiences in Skin Care Clinical Trials
Brief Title: Evaluating Patient Experiences in Skin Care Clinical Studies
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80190623
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Skin Care
Keywords: Skin Care

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrollment in clinical trials usually favors a particular demographic group. But there is limited research available to explain what study attributes affect the completion of these specific demographic groups.

This trial will evaluate the safety and efficacy of new skin care products and treatments. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future skin care studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is able and willing to comply with the treatment/follow-up schedule and requirements
* Patient must provide written informed consent

Exclusion Criteria:

* Women who are pregnant, intend to become pregnant, or are lactating
* Inability to perform regular electronic reporting
* Participants who are vulnerable to any intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational skin care clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a skin care clinical study. | 3 months
Number of skin care study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lichterfeld-Kottner A, El Genedy M, Lahmann N, Blume-Peytavi U, Buscher A, Kottner J. Maintaining skin integrity in the aged: A systematic review. Int J Nurs Stud. 2020 Mar;103:103509. doi: 10.1016/j.ijnurstu.2019.103509. Epub 2019 Dec 23. PMID 31945604
- [Background] Lichterfeld A, Hauss A, Surber C, Peters T, Blume-Peytavi U, Kottner J. Evidence-Based Skin Care: A Systematic Literature Review and the Development of a Basic Skin Care Algorithm. J Wound Ostomy Continence Nurs. 2015 Sep-Oct;42(5):501-24. doi: 10.1097/WON.0000000000000162. PMID 26165590
- [Background] Kottner J, Boronat X, Blume-Peytavi U, Lahmann N, Suhr R. The epidemiology of skin care provided by nurses at home: a multicentre prevalence study. J Adv Nurs. 2015 Mar;71(3):570-80. doi: 10.1111/jan.12517. Epub 2014 Aug 27. PMID 25159337

DOCUMENTS (1):
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT05738018/ICF_000.pdf